CLINICAL TRIAL: NCT02734147
Title: The Efficacy of Intravenous Ascorbic Acid in Patients With Severe Sepsis
Brief Title: High Dose Intravenous Ascorbic Acid in Severe Sepsis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial prematurely terminated due to the loss of funding.
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 603204
Record Dates: First submitted 2016-03-18; First posted 2016-04-12 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose IV ascorbic acid (Active Comparator): Patients will receive 67 mg/kg IV ascorbic acid in 100 ml normal saline over 30 minutes every 8 hours (200 mg/kg/day) for 72 hours.
  Interventions: Drug: Ascorbic Acid
- Placebo (Placebo Comparator): The placebo group will receive 100 ml 0.9% NaCl over 30 minutes every 8 hours for 72 hours.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Ascorbic Acid
  Arms: High dose IV ascorbic acid
Other: Normal Saline
  Arms: Placebo

SUMMARY:
Despite an organized treatment approach outlined in expert-consensus guidelines for sepsis with fluid resuscitation to treat hypovolemia, antibiotics to target the infectious insult, and vasopressors for hypotension, mortality rates for sepsis remain high and the incidence continues to rise, making sepsis the most expensive inpatient disease.

1. Recent research has described the therapeutic benefits associated with ascorbic acid treatment for sepsis.
2. Researchers objectives are to perform a randomized-controlled clinical trial investigating the ability of ascorbic acid(vitamin C) administration to decrease organ dysfunction in severe sepsis. The widespread occurrence of microvascular dysfunction in sepsis leading to tissue hypoxia, mitochondrial dysfunction, and adenosine triphosphate (ATP) depletion, gives rise to organ failure.
3. Patients with organ failure and sepsis (severe sepsis) are at a higher risk of death than patients with organ failure alone. Critically ill patients may have an increased requirement for ascorbic acid in sepsis and these patients frequently have levels below normal. Ascorbic acid administration, has been shown to correlate inversely with organ failure (human literature) and directly with survival (animal studies).

4,5 Intravenous ascorbic acid therapy decreases organ failure by providing a protective effect on several microvascular functions including improving capillary blood flow, decreasing microvascular permeability, and improving arteriolar responsiveness to vasoconstrictors. Defining the utility of novel agents to augment researchers care for severe sepsis is an important task as investigators continue the institutional focus on sepsis care.

ELIGIBILITY:
Inclusion Criteria:

Patients with:

1. A suspected or confirmed infection with an order for intravenous antibiotics or antivirals
2. The presence of acute sepsis-induced organ dysfunction

Definition of organ dysfunction:

1. Arterial hypoxemia [PaO2 /FiO2 < 300]
2. Hypotension [systolic blood pressure (SBP) < 90 mmHg or SBP decrease > 40 mmHg]
3. Lactic acidosis [lactate > 2.5 mmol/L]
4. Acute kidney injury [creatinine >2.0 or urine output < 0.5 ml/kg/hr for >2 hours despite fluid resuscitation]
5. Thrombocytopenia [platelet count < 100,000]
6. Acute coagulopathy [international normalized ratio (INR) > 1.5]
7. Hepatic failure [bilirubin > 2 mg/dL].
8. Predisposition, Infection, Response, and Organ Failure (PIRO) score ≥ 10

Exclusion Criteria:

1. Age < 18 years
2. Pregnancy or breastfeeding
3. Requirement for immediate surgery within the treatment protocol timeframe
4. Inability to obtain written informed consent from subject or surrogate
5. Patient to receive comfort measures only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04-01; Primary Completion 2017-10-08 (Actual); Study Completion 2017-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Arnold, MD, Principal Investigator — Christiana Care Health Services; Jamie Rosini, PharmD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Chrisitana Care Health System-Christiana Hospital, Newark, Delaware, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose IV Ascorbic Acid: Patients will receive 67 mg/kg IV ascorbic acid in 100 ml normal saline over 30 minutes every 8 hours (200 mg/kg/day) for 72 hours.
  Ascorbic Acid
  Participant Started: 12 Participant Completed: 9
- Placebo: The placebo group will receive 100 ml 0.9% NaCl over 30 minutes every 8 hours for 72 hours.
  Normal Saline
  Participant Started: 12 Participant Completed: 11
Period: Overall Study
Arm/Group | High Dose IV Ascorbic Acid | Placebo
Started | 12 | 12
Completed | 9 | 11
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- High Dose IV Ascorbic Acid: Patients will receive 67 mg/kg IV ascorbic acid in 100 ml normal saline over 30 minutes every 8 hours (200 mg/kg/day) for 72 hours.
  Ascorbic Acid
- Placebo: The placebo group will receive 100 ml 0.9% NaCl over 30 minutes every 8 hours for 72 hours.
  Normal Saline
- Total: Total of all reporting groups
Arm/Group | High Dose IV Ascorbic Acid | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (13.6) | 70.2 (14.4) | 68.9 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 7 | 9 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Ascorbic Acid Concentration, Baseline [Mean (Standard Deviation); unit: mg/dL] — Normal Ascorbic Acid Range 0.4-2.0 mg/dL Population: Missing Data
  mg/dL
    number analyzed (Participants) | 11 | 11 | 22
    (all) | 0.3 (0.3) | 0.4 (0.3) | 0.3 (0.3)
Ascorbic Acid Concentrations <0.4 mg/dL, Baseline [Number; unit: percentage of participants] — Normal Ascorbic Acid Range 0.4-2.0 mg/dL Population: Missing data
  percentage of participants
    number analyzed (Participants) | 11 | 11 | 22
    (all) | 72.7 | 36.6 | 68.1
PIRO Score, Baseline [Mean (Standard Deviation); unit: scores on a scale] — PIRO consists of 4 assessments, Predisposition (scored 0-9), Infection (scored 0-4), Response (scored 0-6), and Organ Failure (scored 0-14). The total PIRO score is the sum of all subscores and ranges from 0-33 with higher scores indicating worse health
  scores on a scale | 15.4 (3.9) | 15.9 (4.0) | 15.7 (3.9)
Modified SOFA Score, Baseline [Mean (Standard Deviation); unit: units on a scale] — Sequential Organ Failure Assessment (SOFA) Score included the degree of dysfunction of six organ systems (Respiratory, Cardiovascular, Liver, Renal, Coagulation, Neurologic. A modification of the SOFA includes the exclusion of the Liver function. Total score is reported, minimum score = 0 maximum score = 20. Higher scores indicate greater degree of dysfunction.
  units on a scale | 5.2 (2.5) | 5.0 (2.3) | 5.1 (2.3)
ICU Admission [Count of Participants; unit: Participants] | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified SOFA Score
Description: Sequential Organ Failure Assessment (SOFA) Score included the degree of dysfunction of six organ systems (Respiratory, Cardiovascular, Liver, Renal, Coagulation, Neurologic. A modification of the SOFA includes the exclusion of the Liver function. Total score is reported, minimum score = 0 maximum score = 20. Higher scores indicate greater degree of dysfunction.
Time Frame: Baseline and 72 hours
Population: Data was not available for 3 participants in the treatment group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Dose IV Ascorbic Acid | Placebo
Number analyzed (Participants) | 9 | 12
units on a scale | -1.0 (4.4) | -1.75 (3.0)
Statistical Analysis 1: Comparison: High Dose IV Ascorbic Acid vs Placebo; Test type: Other; p = 0.631, Other

2. Secondary Outcome: Modified SOFA Score
Description: Sequential Organ Failure Assessment (SOFA) Score included the degree of dysfunction of six organ systems (Respiratory, Cardiovascular, Liver, Renal, Coagulation, Neurologic. A modification of the SOFA includes the exclusion of the Liver function. Total score is reported, minimum score = 0 maximum score = 20. Higher scores indicate greater dysfunction.
Time Frame: at 72 Hours
Population: Data was not available for 3 participants in the treatment group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Dose IV Ascorbic Acid | Placebo
Number analyzed (Participants) | 9 | 12
units on a scale | 4.1 (4.8) | 3.3 (3.7)
Statistical Analysis 1: Comparison: High Dose IV Ascorbic Acid vs Placebo; Test type: Other; p = 0.640, Other

3. Secondary Outcome: Ascorbic Acid Concentration at 32 Hours
Description: Ascorbic Acid Concentration Normal Ascorbic Acid Range 0.4-2.0 mg/dL
Time Frame: 32 Hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High Dose IV Ascorbic Acid | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL | 13.8 (10.9) | 0.22 (0.21)
Statistical Analysis 1: Comparison: High Dose IV Ascorbic Acid vs Placebo; Test type: Superiority; p = 0.006, Fisher Exact

4. Secondary Outcome: ICU Length of Stay
Description: ICU Length of Stay in Hours
Time Frame: Length of ICU stay up to 200 hours
Population: Data was not available for 7 participants in both groups.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | High Dose IV Ascorbic Acid | Placebo
Number analyzed (Participants) | 5 | 5
Hours | 29 [6 to 187] | 47 [39 to 144]
Statistical Analysis 1: Comparison: High Dose IV Ascorbic Acid vs Placebo; Test type: Superiority; p = 0.655, Fisher Exact

5. Secondary Outcome: Hospital Length of Stay
Description: From admission until discharge from ICU in days
Time Frame: From ICU admission through ICU discharge, up to 2 weeks
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | High Dose IV Ascorbic Acid | Placebo
Number analyzed (Participants) | 12 | 12
Days | 7 [5 to 9] | 6 [4 to 7]
Statistical Analysis 1: Comparison: High Dose IV Ascorbic Acid vs Placebo; Test type: Superiority; p = 0.133, Fisher Exact

6. Secondary Outcome: Change in PIRO Score
Description: PIRO consists of 4 assessments, Predisposition (scored 0-9), Infection (scored 0-4), Response (scored 0-6), and Organ Failure (scored 0-14) (PIRO). The total PIRO score is the sum of all subscores and ranges from 0-33 with higher scores indicating worse health.
Time Frame: Baseline and 72 hours
Population: Data was not available for 3 participants in the treatment group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Dose IV Ascorbic Acid | Placebo
Number analyzed (Participants) | 9 | 12
units on a scale | -3.7 (3) | -4.5 (3.9)
Statistical Analysis 1: Comparison: High Dose IV Ascorbic Acid vs Placebo; Test type: Other; p = 0.566, Other

7. Secondary Outcome: Percentage of Participants Who Died
Time Frame: From initial hospital admission through discharge, up to 2 weeks.
Measure: Number; unit: Percentage of participants
Arm/Group | High Dose IV Ascorbic Acid | Placebo
Number analyzed (Participants) | 12 | 12
Percentage of participants | 16.7 | 16.7
Statistical Analysis 1: Comparison: High Dose IV Ascorbic Acid vs Placebo; Test type: Superiority; p = 1.0, Chi-squared

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | High Dose IV Ascorbic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 2/12 | 2/12
Serious Adverse Events (participants affected / at risk) | 2/12 | 2/12
Other Adverse Events (participants affected / at risk) | 6/12 | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose IV Ascorbic Acid (N=12) | Placebo (N=12)
Death (General disorders) | 2 | 2
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Short of breath during the 48-72 hour post randomization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose IV Ascorbic Acid (N=12) | Placebo (N=12)
Hypotension (SBP< 90) (Vascular disorders) | 2 (3) | 0 (0)
Tachycardia (HR increase 20 bpm) (Cardiac disorders) | 1 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Other (General disorders) | 4 (8) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT02734147/Prot_SAP_000.pdf